CLINICAL TRIAL: NCT00892346
Title: Phase III Study of Single Autologous Stem Cell Transplantation Followed by Maintenance Therapy as Front-line Treatment for Myeloma
Brief Title: Single Autologous Stem Cell Transplantation Followed by Maintenance Therapy as Front-line Treatment for Myeloma
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: No avaliability of melphlan in mainland China
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHOPES-myeloma09
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: autologous hematopoietic stem cell transplantation; maintenance
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single ASCT with Thalidomide maintenance (Experimental): Single ASCT followed by Thalidomide maintenance:
  1. patients recieved 4-6 cycles of standard VAD chemotherapy or Thalidomide/dexamethasone as induction therapy
  2. CTX+G-SCF mobilization to collecetd PBSC
  3. Patiens recieved Mel 200 as conditioning followed by Thalidomide 100mg maintenance
  Interventions: Procedure: Single ASCT with Thalidomide maintenance

INTERVENTIONS:
Procedure: Single ASCT with Thalidomide maintenance — Single ASCT with Thalidomide maintenance:
  1. Single Autologous Stem Cell Transplantation: conditioning with Melphalan 200mg/m2 (iv)
  2. Thalidomide maintenance: starting from D60 after transplantation at 100-200mg daily (Oral)
  Other Names: multiple myeloma; melphalan; thalidomie

SUMMARY:
The clinical trial is to evaluate the efficacy of single autologous hematopoietic stem cell transplantation with standard conditioning of melphalan 200 mg/m2 followed by thalidomide maintenance in patients with newly-diagnosed myeloma after receiving 4-6 cycles of induction chemotherapy consisting of vincristin,adriamycin and dexamethasone (VAD) or thalidomide/dexamethasone between 18 to 65 years.

DETAILED DESCRIPTION:
This is an open label clinical trial to evaluate the efficacy of single autologous hematopoietic stem cell transplantation in newly diagnosed multiple myeloma patients. All patients will receive 4-6 cycles of induction therapy which includes VAD chemotherapy (vincristin, adriamycin and dexamethasone) or thalidomide/dexamethasone. After peripheral hematopoietic stem cell mobilization and apheresis, patients will receive a standard conditioning with melphalan 200mg/m2 followed by thalidomide maintenance therapy at 100-200mg orally daily starting from D+60 till disease progression or untolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between age 18-65 with newly diagnosed Multiple Myeloma for whom stem cell transplantation is considered appropriate
* Measurable serum and/or urinary paraprotein
* European Cooperative Oncology Group performance status 0-3
* Serum bilirubin < 1.5x the upper limit of normal (ULN)
* Serum alanine transaminase (ALT)/aspartate transaminase values < 2.5 x ULN
* Subjects (or their legally acceptable representatives) must signed an informed consent document indicating that they understanding the purpose of and procedures required for the study and are willing to participate in the study

Exclusion criteria:

* Woman of child bearing potential
* Non-secretory MM
* Serum creatinine > 400 Micromol/l after initial resuscitation
* patients with previous Grade 2-4 peripheral neuropathy
* Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, uncontrolled angina, clinically significant pericardial disease, or III-IV heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
response rate: CR/nCR/VGPR | 6 months after auto-PBSCT

SECONDARY OUTCOMES:
overall survival | 3 years
progression free survival | 3 years
toxicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, M.D., Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Rui Jin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang JE, Juckett MB, Callander NS, Kahl BS, Gangnon RE, Mitchell TL, Longo WL. Thalidomide maintenance following high-dose melphalan with autologous stem cell support in myeloma. Clin Lymphoma Myeloma. 2008 Jun;8(3):153-8. doi: 10.3816/CLM.2008.n.018. PMID 18650178
- [Background] Abdelkefi A, Ladeb S, Torjman L, Othman TB, Lakhal A, Romdhane NB, Omri HE, Elloumi M, Belaaj H, Jeddi R, Aissaoui L, Ksouri H, Hassen AB, Msadek F, Saad A, Hsairi M, Boukef K, Amouri A, Louzir H, Dellagi K, Abdeladhim AB; Tunisian Multiple Myeloma Study Group. Single autologous stem-cell transplantation followed by maintenance therapy with thalidomide is superior to double autologous transplantation in multiple myeloma: results of a multicenter randomized clinical trial. Blood. 2008 Feb 15;111(4):1805-10. doi: 10.1182/blood-2007-07-101212. Epub 2007 Sep 17. PMID 17875806 (Retraction: PMID 19520824 Abdelkefi A, Ladeb S, Torjman L, Ben Othman T, Lakhal A, Ben Romdhane N, Elloumi M, Jeddi R, Aissaouï L, Ben Hassen A, Msadek F, Saad A, Hsaïri M. Blood. 2009 Jun 11;113(24):6265)
- [Background] Harousseau JL, Moreau P. Evolving role of stem cell transplantation in multiple myeloma. Clin Lymphoma Myeloma. 2005 Sep;6(2):89-95. doi: 10.3816/CLM.2005.n.034. PMID 16231846
- [Background] Spencer A, Prince HM, Roberts AW, Prosser IW, Bradstock KF, Coyle L, Gill DS, Horvath N, Reynolds J, Kennedy N. Consolidation therapy with low-dose thalidomide and prednisolone prolongs the survival of multiple myeloma patients undergoing a single autologous stem-cell transplantation procedure. J Clin Oncol. 2009 Apr 10;27(11):1788-93. doi: 10.1200/JCO.2008.18.8573. Epub 2009 Mar 9. PMID 19273705
- [Background] Kumar A, Kharfan-Dabaja MA, Glasmacher A, Djulbegovic B. Tandem versus single autologous hematopoietic cell transplantation for the treatment of multiple myeloma: a systematic review and meta-analysis. J Natl Cancer Inst. 2009 Jan 21;101(2):100-6. doi: 10.1093/jnci/djn439. Epub 2009 Jan 13. PMID 19141779